CLINICAL TRIAL: NCT03329118
Title: Drug Interaction Study of Henagliflozin and Simvastatin in Healthy Volunteers
Brief Title: Drug-drug Interaction Between Simvastatin and SHR3824
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3824-111
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
Keywords: SHR3824,simvastatin, drug-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin; Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR3824 1Omg,Simavastatin 40mg (Experimental): two 20mg tablets of simvastatin once daily on Day 1 followed by one 10mg tablet of SHR3824 once daily on Day 4,5,6,7,followed by two 20mg tablets of simvastatin and one 10mg tablet of SHR3824 on Day 8.
  Interventions: Drug: SHR3824, Simvastatin

INTERVENTIONS:
Drug: SHR3824, Simvastatin — two 20mg tablets of simvastatin once daily on Day 1 followed by one 10mg tablet of SHR3824 once daily on Day 4,5,6,7,followed by two 20mg tablets of simvastatin and one 10mg tablet of SHR3824 on Day 8.

SUMMARY:
the purpose of thr study is to investigate the potential interation between multiple oral doses of SHR3824 and single oral dose of Simvastatin in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 19 and 26 kg/m2

Exclusion Criteria:

* History of hypoglycemia
* History of urinary tract infections,or genital infections
* History of current clinically significant medical illness as determined by the Investigator
* Known allergy to SHR3824 or Simvastatin or any of the excipients of the formulation of SHR3824 or Simvastatin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-11-24 (Estimated); Primary Completion 2017-12-04 (Estimated); Study Completion 2017-12-08 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SHR3824 | At protocol-specified times up to Day 7 and Day 8
  Cmax (a measure of the body's exposure to SHR3824) will be compared before and after coadministration with Simvastatin .
The area under the plasma concentration-time curve (AUC) of SHR3824 | At protocol-specified times up to Day 7 and Day 8
  AUC(a measure of the body's exposure to SHR3824) will be compared before and after coadministration with Simvastatin .
The area under the plasma concentration-time curve (AUC) of Simvastatin and simavastatin acid . | At protocol-specified times up to Day 1 and Day 8
  AUC(a measure of the body's exposure to simvastatin and simavastatin acid) will be compared before and after coadministration with SHR3824 .
The maximum plasma concentration (Cmax) of simvastatin and simavastatin acid. | At protocol-specified times up to Day 1 and Day 8
  Cmax (a measure of the body's exposure to simvastatin and simavastatin acid) will be compared before and after coadministration with Simvastatin .
The number of volunteers with adverse events as a measure of safety and tolerability. | up to day 15